CLINICAL TRIAL: NCT04408703
Title: PRognOstiC valuE of rEd Density in Ulcerative Colitis: PROCEED-UC STUDY
Brief Title: PRognOstiC valuE of rEd Density in Ulcerative Colitis
Acronym: PROCEED-UC
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Sapporo Medical University (Other); Imelda GI Clinical Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: s63012
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2020-05

CONDITIONS: Ulcerative Colitis
Keywords: Endoscopy; Artificial intelligence; Image analysis; Precision medicine; Inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum albumin, faecal calprotectin, C-reactive protein, thrombocytosis and haemoglobin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ulcerative colitis in clinical remission: Clinical remission with SCCAI <3 at baseline and stable remission for the last 3 months
  Interventions: Diagnostic Test: Red Density

INTERVENTIONS:
Diagnostic Test: Red Density — Image analysis of endoscopic images in patients with ulcerative colitis

SUMMARY:
Observational prospective multicenter study: baseline assessement of the disease activity by an automated endoscopic tool and follow up of 52 weeks to evaluate sustained clinical remission.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of UC for at least 3 months
* Clinical remission with SCCAI <3 at baseline and stable remission for the last 3 months
* Ability to give informed consent by the patient or legal representative in case of minority.

Exclusion Criteria:

* Any contraindication for sigmoidoscopy or undergoing biopsies of the rectosigmoid.
* Uncontrolled coagulopathy.
* Any planned change in UC related treatment (both escalation and de-escalation) after the baseline endoscopy
* Planned UC related surgery
* Previous subtotal or total colectomy
* Short bowel, ileostomy or colostomy
* Pregnancy at baseline
* Age younger than 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ulcerative colitis in clinical remission
Sampling Method: Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
sustained clinical remission | week 52
  Number of patients with sustained clinical remission at week 52, defined as simple clinical colitis activity index (SCCAI) <3 AND no need for initiation of new treatment, escalation of therapy, UC related hospitalization or colectomy correlated to the RD score at baseline.

SECONDARY OUTCOMES:
endoscopic remission Mayo | week 52
  Number of patients with Mayo endoscopic subscore of 0 after 52 weeks correlated to the RD score at baseline.
endoscopic remission UCEIS | week 52
  Number of patients with UCEIS of 0 after 52 weeks correlated to the RD score at baseline.

OTHER OUTCOMES:
correlation biomarker | week 52
  Correlation between RD scores and fecal calprotectin, C-reactive protein (CRP), platelet count and haemoglobin at any point in the study.
correlation histological score | week 52
  Correlation between RD scores and Geboes histological score, the Nancy and the Robarts histological index at any point in the study.
correlation endoscopic score | week 52
  Correlation between RD scores and Mayo endoscopic subscore and UCEIS at any point in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Raf Bisschops, MD PhD, Principal Investigator — UZ Leuven; Peter Bossuyt, MD, Principal Investigator — UZ Leuven
Locations (2):
- Belgium (2):
  - Imelda GI clinical research center, Bonheiden
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bossuyt P, Nakase H, Vermeire S, de Hertogh G, Eelbode T, Ferrante M, Hasegawa T, Willekens H, Ikemoto Y, Makino T, Bisschops R. Automatic, computer-aided determination of endoscopic and histological inflammation in patients with mild to moderate ulcerative colitis based on red density. Gut. 2020 Oct;69(10):1778-1786. doi: 10.1136/gutjnl-2019-320056. Epub 2020 Jan 8. PMID 31915237